CLINICAL TRIAL: NCT00781209
Title: A Phase II Trial Evaluating the Role of Posterior Fossa Irradiation (PFI) Plus Stereotactic Radiosurgery (SRS) for Cerebellar Metastases
Brief Title: The Role of Posterior Fossa Irradiation (PFI) Plus Stereotactic Radiosurgery (SRS) for Cerebellar Metastases
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Prof. Ben Corn, Radiotherapy Department, TASMC
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TASMC - 08 - BC - 270 - CTIL
Record Dates: First submitted 2008-10-26; First posted 2008-10-28 (Estimated); Last update posted 2008-10-28 (Estimated); Status verified 2008-10

CONDITIONS: Neoplasm Metastasis
Keywords: irradiation; stereotactic radiosurgery; posterior fossa; cerebellar metastases
MeSH Terms: conditions — Neoplasm Metastasis | interventions — Radiation; Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Exp (Experimental): Posterior Fossa Irradiation 37.5 Gy in 2.5 Gy fractions+Radiosurgical boost; Follow up:Contrast enhanced MRI & Mini Mental Status Examination
  Interventions: Procedure: Irradiation plus Stereotactic Radiosurgery

INTERVENTIONS:
Procedure: Irradiation plus Stereotactic Radiosurgery — Posterior Fossa Irradiation-total dose of 37.5 Gy in 2.5 Gy fractions administered via conformal beams.
  Radiosurgical boost-total dose administered to each lesion will be titrated to the size of the metastatic focus as follows:
  Maximum Tumor Diameter:<2.0 cm; Assigned Dose:24 Gy. Maximum Tumor Diameter:2.1-3.0 cm;Assigned Dose:18 Gy. Maximum Tumor Diameter:3.1-4.0 cm;Assigned Dose:15 Gy.

SUMMARY:
The aggregate of data pertaining to brain metastases suggests that optimal results are achievable with a 2-pronged approach that addresses both the specific focus (with surgery or radiosurgery) and the surrounding brain parenchymal tissue that may harbor micrometastases. Patterns of failure following treatment of metastases that arise in the posterior fossa have not been reliably defined. Although most would agree that radiosurgery alone is not sufficient treatment for focal metastases in the cerebellum, it may be possible to deliver less than WBI as an "expanded port" beyond the SRS volume.

The current study acknowledges that at least two therapeutic modalities are requisite for patients with cerebellar metastases but hypothesizes that it is unnecessary to extend the treatment of ostensibly uninvolved brain tissue beyond the limits of the posterior fossa. In so doing, it is hoped that the putative advantage derived from foregoing whole brain irradiation (e.g., reduction in neurocognitive impairment) will not be at the expense of excessive surpratentorial failure.

DETAILED DESCRIPTION:
SCHEMA:

* Posterior Fossa Irradiation as defined by diagnostic MRI and CT simulation.
* 37.5 Gy in 2.5 Gy fractions administered via conformal beams.
* Radiosurgical boost (with dose titrated to parameters of RTOG 9005).
* Contrast enhanced MRI will be obtained at baseline and then at 3, 6, and 12 months following completion of posterior fossa irradiation.
* The Mini Mental Status Examination will be used to evaluate global cognitive function at baseline and then at 3, 6, and 12 months following completion of posterior fossa irradiation.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed malignant disease
* All primary tumors exclusive of:

  * Small cell lung cancer
  * Renal cell cancer (hypernephroma)
  * Melanoma
  * Sarcoma
* 1-3 intraparenchymal metastases
* Age ≥18 years
* RPA(14) 1 or 2
* Patients who have undergone resection are eligible provided residual disease is evident on imaging
* No clinical or radiographic evidence of progression of extracranial disease in month prior to enrollment on study.

Exclusion Criteria:

* Major psychiatric illness
* Lesions in brainstem, midbrain, pons, medulla
* Patient who have undergone complete resection of all known infratentorial disease
* Patients with leptomeningeal metastases
* Patients with hepatic metastases
* Patients with metastases from the following primary tumors are ineligible: Small Cell Lung Cancer; rena Cell Carcinoma; Melanoma; Sarcoma
* Previous cranial irradiation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2008-10; Primary Completion 2009-10 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
To determine tumor control rates in the brain following posterior fossa irradiation of patients with cerebellar metastases. | 1 year

SECONDARY OUTCOMES:
To establish levels of neurocognitive performance following posterior fossa irradiation of patients with cerebellar metastases. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Ben Corn, Prof., Principal Investigator — Radiotherapy Department, TASMC
Locations (1):
- Radiotherapy Department, TASMC, Tel Aviv, Israel